CLINICAL TRIAL: NCT01473459
Title: Comparison Between Two Fertility Protocols in Obese Polycystic Ovary Syndrome
Brief Title: Comparison Between Two Fertility Protocols in Obese Polycystic Ovary Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0078-11-HYMC
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Obese; Infertility; Polycystic Ovary Syndrome
Keywords: best fertility protocol; (BMI > 30); women; PCOS
MeSH Terms: conditions — Obesity; Infertility; Polycystic Ovary Syndrome | interventions — Intravital Microscopy; Therapeutics; Fertilization in Vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVM Treatment (Active Comparator)
  Interventions: Procedure: IVM (In Vitro Maturation) Treatment
- Antagonist Protocol (Active Comparator)
  Interventions: Procedure: IVF (In Vitro Fertilization) Antagonist Protocol

INTERVENTIONS:
Procedure: IVM (In Vitro Maturation) Treatment — There will be no gonadotropin stimulation. There will be ovum pickup from antral follicles of immature oocyte which will be matured in the lab and fertilized by intracytoplasmic sperm injection (ICSI). Embryo transfer will take place on days 2 or 3.
  Other Names: IVM
  Arms: IVM Treatment
Procedure: IVF (In Vitro Fertilization) Antagonist Protocol — The first stage of the treatment will be stimulation with gonadotropins. Next GNRH Antagonist will be added. Ovulation induction will be performed with GNRH agonist. After ovulation there will be ovum pickup and fertilization in the lab. Embryo transfer will take place on days 2 or 3.
  Other Names: IVF - antagonist protocol
  Arms: Antagonist Protocol

SUMMARY:
The purpose of this study is to compare two fertility protocols in obese women with Polycystic Ovarian Syndrome who are candidates for In Vitro Fertilization (IVF). These protocols carry less risk of ovarian hyperstimulation syndrome which these women may experience.

DETAILED DESCRIPTION:
The purpose of this study is to compare two fertility protocols in obese women with Polycystic Ovarian Syndrome who are candidates for In Vitro Fertilization (IVF). These protocols carry less risk of ovarian hyperstimulation syndrome which these women may experience.The patients in the IVM group will not be exposeD to gonadotropin treatment for controlled ovarian hyperstimulation. In the antagonist group we will use GnRH agonist to induce ovulation which may reduce the risk for ovarian hyperstimulation.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* PCOS
* Failure of COH treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Fertility results | One year

CONTACTS AND LOCATIONS:
Overall Officials: Tal Shavit, M.D, Principal Investigator — IVF unit Hillel-Yaffe medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel